CLINICAL TRIAL: NCT06288620
Title: A Prospective, Open-label, Single-arm Phase II Clinical Study to Evaluate the Efficacy and Safety of Microwave Ablation in the Treatment of Early-stage Unifocal Invasive Breast Cancer
Brief Title: Microwave Ablation in the Treatment of Early-stage Unifocal Invasive Breast Cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MA-EBC-II-024
Record Dates: First submitted 2024-02-25; First posted 2024-03-01 (Actual); Last update posted 2024-03-01 (Actual); Status verified 2024-02

CONDITIONS: Breast Cancer
Keywords: Ablation
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Microwave Ablation (Experimental): Preoperative US-guided microwave ablation of breast cancer
  Interventions: Procedure: Microwave Ablation

INTERVENTIONS:
Procedure: Microwave Ablation — Preoperative US-guided microwave ablation of breast cancer

SUMMARY:
Microwave Ablative (MWA) therapy, as a minimally invasive thermal therapy, has been attempted to treat breast cancer of small lesions . However, the optimal indications for MWA in the treatment of breast cancer is unknown. This prospective, open-label, single-arm phase II clinical study was conducted to evaluate the efficacy and safety of MWA in the treatment of early-stage unifocal invasive breast cancer, and to explore the immune activating effect.

ELIGIBILITY:
Inclusion Criteria:

1. female patients aged 18-70 years;
2. patients with newly diagnosed invasive breast cancer confirmed by core needle biopsy;
3. the tumor smaller than 2cm in greatest diameter confirmed by US (ultrasonography), breast X-ray and breast MRI (contrast-enhanced magnetic resonance image ) were performed at the same time, and the difference of the largest diameter between breast US and MRI was less than 0.5 cm;
4. the single tumor without other suspicious lesions (BI-RADS (the Breast Imaging Recording and Data System) score ≥4) evaluated by breast US, X-ray and MRI;
5. the tumor without adhesion to chest wall, nipple or skin;
6. patients without distant metastasis;
7. Karnofsky performance status greater than 70%.

Exclusion Criteria:

1. multicentric or multifocal breast tumor;
2. the tumor located on nipple and areola area;
3. signs of extensive intraductal carcinoma on imaging examination (diffuse malignant calcification on breast X-ray or segmental distribution, non-mass enhancement, ductal or linear enhancement > 2.5 cm on MRI);
4. extensive intraductal component in invasive cancer (more than 50% of the tumor volume) confirmed by pathology;
5. invasive lobular carcinoma, metaplastic carcinoma or carcinoma with sclerosing adenosis;
6. patients who were pregnant or breastfeeding;
7. patients with evidence of coagulopathy, chronic liver diseases or renal failure;
8. patients with previous treatment including chemotherapy, targeted drug therapy, or local radiation therapy, etc;
9. patients with substance abuse, or mental or psychological disorders that may interfere with study compliance;
10. any condition that is unstable or likely to compromise the patient's safety and compliance;
11. patients enrolled in other clinical trials;
12. diseases or symptoms that other investigators consider unsuitable for participation.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 77 (Estimated)
Dates: Start 2024-02-25 (Actual); Primary Completion 2025-05-10 (Estimated); Study Completion 2025-05-30 (Estimated)

PRIMARY OUTCOMES:
Complete ablation rate | 1 day
  The proportion of patients with complete ablation was calculated for all patients. Complete ablation was defined as: tissue section at the ablation margin that was negative by histochemical staining.

SECONDARY OUTCOMES:
Safety of microwave ablation | 10 days
  Safety measured by occurrence of study related adverse effects defined by NCI CTCAE 5.0

CONTACTS AND LOCATIONS:
Locations (1):
- the First Affiliated Hospital of Nanjing Medical University, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Yes
Available from the corresponding author upon reasonable request
Supporting Information: Study Protocol